CLINICAL TRIAL: NCT07090122
Title: Radiofrequency Ablation/Bone Augmentation + Radiotherapy vs Radiotherapy Alone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-2023-32509
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Spine Metastases; Bone Pain
Keywords: Radiofrequency ablation (RFA); Bone augmentation (BA); Radiotherapy (RT); Metastatic disease of the spine
MeSH Terms: interventions — Radiofrequency Ablation; Radiotherapy

STUDY DESIGN:
Intervention Model Description: single-center, randomized 2 arm controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation and bone augmentation with radiotherapy (Active Comparator): Radiofrequency-generated heat to eradicate cancer cells, followed by the application of a bone-stabilizing agent to offer both tumor control and structural reinforcement. Radiotherapy (RT) uses high-energy radiation to target and destroy cancer cells, providing notable pain relief and potentially reducing tumor size
  Interventions: Procedure: Radiofrequency ablation and bone augmentation with radiotherapy
- Radiotherapy alone (Placebo Comparator): ONLY uses high-energy radiation to target and destroy cancer cells, providing notable pain relief and potentially reducing tumor size
  Interventions: Procedure: Radiotherapy alone

INTERVENTIONS:
Procedure: Radiofrequency ablation and bone augmentation with radiotherapy — employs radiofrequency-generated heat to eradicate cancer cells, followed by the application of a bone-stabilizing agent
  Arms: Radiofrequency ablation and bone augmentation with radiotherapy
Procedure: Radiotherapy alone — High-energy radiation
  Arms: Radiotherapy alone

SUMMARY:
This is a single-center, randomized controlled pilot study of radiofrequency ablation and bone augmentation (RFA/BA) plus radiotherapy (RT) vs. RT alone in patients with metastatic T5-L5 disease of the spine. Patients will be randomized 2:1 to receive either one treatment of RFA/BA plus RT or RT to evaluate the occurrence of skeletal-related events. Skeletal-related events (SREs) are defined as new clinical or radiologic evidence of pathologic fracture, spinal cord or nerve root compression, pain or instability, and/or necessity for additional local intervention (i.e. surgery, repeat RFA/BA or RT) due to persistent or progressive symptoms. Post-treatment follow-up for SREs are assessed at 1, 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic T5-L5 disease of the spine (with up to two levels) as detected by any imaging study.
* Have either associated bone pain or cross-sectional imaging characteristics that are predictors of SRE.
* Age 18 years of age or older at the time of consent.
* Have adequate organ function confirmed by the following laboratory values obtained within 14 days prior to study enrollment defined as:

  1. absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  2. platelets ≥ 50 × 109/L
  3. hemoglobin ≥ 10 g/dL, independent of transfusion ≤14 days of screening
  4. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); if liver metastases, then ≤ 5 × ULN
  5. total bilirubin ≤ 1.5 × ULN; < 2 × ULN if hyperbilirubinemia is due to Gilbert's syndrome
  6. serum albumin ≥ 30 g/L (3.0 g/dL)
  7. serum creatinine ≤ 1.5 x ULN; OR estimated glomerular filtration rate (GFR) ≥ 45 mL/min using the Cockcroft Gault formula
* Persons of childbearing potential (POCB) or with partners of childbearing potential must be willing to use contraception during study treatment and 6 months after study treatment.
* Persons are considered to be of childbearing potential unless one or the following applies:

  1. Is postmenopausal, defined as no menses for at least 12 months without an alternative medical cause
  2. Considered permanently sterile. Permanent sterilization includes hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy
* Voluntary written consent prior to the performance of any research related activity

Exclusion Criteria:

* Pregnant or breastfeeding.
* Clinical or radiologic evidence of epidural spinal cord compression or radicular pain.
* Prior radiation therapy to the target lesion.
* Candidates for spine stabilization surgery.
* The target lesion(s) is deemed ineligible for RFA/BA (e.g. unstable existing fractures/impending fractures, involvement of the posterior elements, retropulsion, spinal canal narrowing, neuroforaminal narrowing, uncontrolled bleeding diathesis, active infection anywhere in the body, or purely blastic tumor). Note: Mixed lytic/blastic tumors are eligible.
* The target lesion(s) size or location is beyond RFAs ability to safely perform, at the physician's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-01-13 (Estimated); Study Completion 2028-06-13 (Estimated)

PRIMARY OUTCOMES:
Skeletal-related event (SREs) outcomes at 1 month | Month 1
  Skeletal-related events are defined as new clinical or radiologic evidence of pathologic fracture, spinal cord or nerve root compression, pain or instability, and/or necessity for additional local intervention (i.e. surgery, repeat RFA/BA or RT) due to persistent or progressive symptoms.
Skeletal-related event (SREs) outcomes at 3 months | Month 3
  Skeletal-related events are defined as new clinical or radiologic evidence of pathologic fracture, spinal cord or nerve root compression, pain or instability, and/or necessity for additional local intervention (i.e. surgery, repeat RFA/BA or RT) due to persistent or progressive symptoms.
Skeletal-related event (SREs) outcomes at 6 months | Month 6
  Skeletal-related events are defined as new clinical or radiologic evidence of pathologic fracture, spinal cord or nerve root compression, pain or instability, and/or necessity for additional local intervention (i.e. surgery, repeat RFA/BA or RT) due to persistent or progressive symptoms.
Skeletal-related event (SREs) outcomes at 12 months | Month 12
  Skeletal-related events are defined as new clinical or radiologic evidence of pathologic fracture, spinal cord or nerve root compression, pain or instability, and/or necessity for additional local intervention (i.e. surgery, repeat RFA/BA or RT) due to persistent or progressive symptoms.
Skeletal-related event (SREs) outcomes at 24 months | Month 24
  Skeletal-related events are defined as new clinical or radiologic evidence of pathologic fracture, spinal cord or nerve root compression, pain or instability, and/or necessity for additional local intervention (i.e. surgery, repeat RFA/BA or RT) due to persistent or progressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Talaie, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No